CLINICAL TRIAL: NCT02556047
Title: A Clinical Investigation to Evaluate the Safety and Performance of Two Star Intradermal Safety Device (IDSD) Syringes in Healthy Adult Volunteers
Brief Title: Evaluation of the Safety & Performance of 2 Intradermal Safety Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CRC332
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Syringe

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injections (Other): * Two injections of 0.1 ml sterile saline per injection using Star intradermal safety device 1.2mm needle length
  * Two injections of 0.1 ml sterile saline per injection using Star intradermal safety device 1.5mm needle length
  * Two injections of 0.1 ml saline per subject using Mantoux technique by N&S
  Interventions: Device: Star Intradermal Safety Device

INTERVENTIONS:
Device: Star Intradermal Safety Device — Star Intradermal Safety Device 1.2mm needle length, Star Intradermal Safety Device 1.5mm needle length, Mantoux technique by N&S

SUMMARY:
Several vaccinations are administered by the intradermal (ID) method where the vaccine is injected between layers of skin. The current technique required to do this can be difficult to learn and perform accurately, is slower to deliver than subcutaneous or intramuscular injections, and there is a risk that the injection will be given to too-deep skin layers or to underlying tissues, which might change the immune response. There is increasing interest in using ID administration for vaccines as it may be possible to achieve the same immune response with a smaller dose of vaccine. This could increase access to vaccines that are expensive or are only available in small quantities and therefore could have global health benefit for vaccine programs for diseases such as yellow fever and polio.

Because of the potential global-health benefits of being able to give ID injections of vaccines easily, quickly and with relatively little training or experience, several novel devices are currently being developed to allow easy ID administration. Star Syringe have developed two novel intradermal safety devices that differ only in the length of the needle used. The current study will assess how the two new devices perform, compared to the traditional Mantoux test, using injections of saline into the upper arm. Twenty volunteers (18-60 years, male and female) will be recruited and attend a screening visit (1), an injection visit (2a) and have a follow up telephone call (2b). At the injection visit they will receive 3 injections in each arm (Mantoux and 2 device injections) and measurements will be performed.

A subset of volunteers will be invited back to attend an additional visit (3a) which will be a repeat of visit 2 but with an ultrasound image taken of each injection site. There will be a follow up telephone call 24 hours later (3b).

DETAILED DESCRIPTION:
Volunteers will be asked to attend Surrey CRC for two visits with a follow up telephone call. A subset of volunteers will be aske to attend an additional visit and follow up call.

Visit 1 - Screening Visit (Day - 28 to -1) Visit 1 will take place up to 28 days prior to the injections being administered (Visit 2). At this visit consent will be taken and the following procedures performed: demography, medical history and concomitant medication, vital signs (blood pressure, heart rate, oral temperature), symptoms-directed physical examination including assessment of deltoid area, measurement of height and weight, blood sample taken for haematology and coagulation screen, completion of a medical health questionnaire. Inclusion/exclusion criteria will be assessed and volunteers that continue to be eligible will be invited back to attend Visit 2a.

Visit 2a - Injection (Day 0) At Visit 2a, continuing eligibility will be assessed and both adverse events and concomitant medication will be recorded. Vital signs will be measured and if the volunteer is still eligible then they will be randomised onto the study.

The volunteer will receive a total of 6 injections, 3 in each upper arm. In each arm there will be one Mantoux injection and 2 device injections (the same device or different). In total they will receive 2 Mantoux injections and 2 injections from each device. To maintain the blind of the study the volunteers will be asked to wear a blindfold during the injections. After each injection a number of measurements will be performed including assessing wheal size and wetness at the injection site as well as subjectively assessing pain. In addition the devices will be weighed before and after use.

Following the injections, vital signs will be recorded again and volunteers will be discharged and provided with a diary card to complete over the following 24 hours. They should record side effects and any medications taken, including over the counter medications as well as any skin reactions.

Visit 2b - Mandatory Follow Up telephone call (Day 1) The volunteer will be telephoned by a member of the study team 24 hours after the injection visit and both adverse events and concomitant medication will be recorded. Volunteers will be asked to return their diary cards to the CRC in the mail.

A subset of volunteers will be invited back to attend Visits 3a and 3b.

Visit 3a - Injection (Within days 7 to 28) At Visit 3a, continuing eligibility will be assessed and both adverse events and concomitant medication will be recorded. Vital signs will be measured and if the volunteer is still eligible then they will be randomised onto the study.

The volunteer will receive a total of 6 injections, 3 in each upper arm. In each arm there will be one Mantoux injection and 2 device injections (the same device or different). In total they will receive 2 Mantoux injections and 2 injections from each device. To maintain the blind of the study the volunteers will be asked to wear a blindfold during the injections. After each injection a number of measurements will be performed including assessing wheal size and wetness at the injection site as well as subjectively assessing pain. At this visit, ultrasound echography will be performed for each injection site. In addition the devices will be weighed before and after use.

Following the injections, vital signs will be recorded again and volunteers will be discharged and provided with a diary card to complete over the following 24 hours. They should record side effects and any medications taken, including over the counter medications as well as any skin reactions.

Visit 3b - Follow Up telephone call (24 h after Visit 3a) The volunteer will be telephoned by a member of the study team 24 hours after the injection visit and both adverse events and concomitant medication will be recorded. Volunteers will be asked to return their diary cards to the CRC in the mail.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers aged 18 to 60 years inclusive. Attempts will be made to achieve an equal gender ratio through appropriate screening procedures, but a failure to do so will not preclude analysis of the final data set.
2. The volunteer is, in the opinion of the investigator, healthy on the basis of self-reported medical history, vital signs, a physical examination (including the skin overlying the deltoids of the upper arms), and the results of routine haematology and coagulation laboratory tests, with no active disease process that could interfere with the study endpoints.
3. Body Mass Index ≥18.5 and <29.5.
4. The volunteer is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
5. The volunteer has signed the ICF and is willing to comply with study procedures.
6. Available for follow-up for the duration of the study.

Exclusion Criteria:

* 1. Clinically significant psychiatric, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological (particularly myasthenia gravis), immunological, or haematological disease or abnormality, as determined by the study physician, which might interfere with consenting or self-recording of safety events.

  2. Presence of large or dark tattoos or other marking or abnormal variation in skin pigmentation in the area of the deltoids that would preclude measurement of six injection site wheals.

  3. Acute, self-reported needle phobia. 4. Regular use of anti-coagulant medication, non-steroidal anti-inflammatory drugs, topical or oral steroids, anti-histamines and opiates for longer than six months.

  5. Pregnant or lactating at any point during the study from screening to final follow up.

  6. Any condition that, in the investigator's opinion, compromises the volunteers' ability to meet protocol requirements or to complete the study.

  7. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

  8. Dermatological and other conditions likely to cause excessive soreness, bleeding or pain at the site of injection or subsequent scarring; these might include hyperkeratosis and bleeding disorders.

  9. Peripheral neuropathy, which might interfere with pain perception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Diameter of wheal following each injection | Within 2 minutes
  To obtain data on wheal size for two versions of an investigational intradermal safety device and compare this to the 'gold-standard' of the Mantoux technique with needle and syringe (referred to as Mantoux N&S)

SECONDARY OUTCOMES:
Volume of fluid on skin following each injection | Within 1 minute
  To obtain data on 'wetness' of injection
Weight of syringes pre filling | Within 4 hours
  To obtain data on pre- and post-injection weight of injectate in the injection devices.
Weight of syringes post filling | Within 2 hours
  To obtain data on pre- and post-injection weight of injectate in the injection devices.
Weight of syringes post injections | Within 2 hours
  To obtain data on pre- and post-injection weight of injectate in the injection devices.
Number of adverse events recorded | Within 24 hours
  Local and systemic safety events recorded. Local safety events will be skin reactivity (redness, hardness, swelling).
Visual Analogue Score for Pain | Within 2 minutes of injections at visit 2a and visit 3a
  Intensity of and comparative perceived pain during injection.
Least painful injection | Within 4 minutes
  Following 3 injections on one arm the participant will be asked which was the least painful injection.
Most painful injection | Within 4 minutes
  Following 3 injections on one arm the participant will be asked which was the most painful injection.
Ease of Use Questionnaire | Within 1 week
  Limited qualitative data on ease of use from the research nurses.

OTHER OUTCOMES:
Depth of dermis | Within 10 mins
  Ultrasound echography of the wheal depth and diameter for two versions of an investigational intradermal safety device, compared with Mantoux N&S
Thickness of dermis | Within 10 mins
  Ultrasound echography of the wheal depth and diameter for two versions of an investigational intradermal safety device, compared with Mantoux N&S

CONTACTS AND LOCATIONS:
Overall Officials: David Lewis, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom